CLINICAL TRIAL: NCT01952990
Title: A Single-Center, Study Evaluating The Pharmacokinetics Of Tetracaine, Para-Butylaminobenzoic Acid, And Oxymetazoline After Intranasal Administration Of Kovacaine Mist To Healthy Pediatric Subjects
Brief Title: Safety and Pharmacokinetics of Kovacaine Nasal Spray in Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Triligent International (Industry); Analytical Bio-Chemistry Laboratories, Inc. (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR 2-07
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Anesthesia
Keywords: Pharmacokinetic
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kovacaine Mist (Experimental): Tetracaine HCl 3% and Oxymetazoline HCl 0.05% - Total dose is based on weight. Subjects weighing 10 to <20 kg will receive 1 intranasal spray of 100 μL. Subjects weighing 20 to <40 kg will receive 2 intranasal sprays of 100 μL (total dose 200 μL.
  Subjects weighing 40 kg or more will receive 2 intranasal sprays of 200 μL (total dose 400 μL).
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%

INTERVENTIONS:
Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% — 1 spray device is 0.2mL (200 μL) in volume and contains 6mg Tetracaine HCl 3% and 0.1mg Oxymetazoline HCl. Subjects receiving the 100 μL dose will receive half of the contents of one device using a dose divider. Subjects receiving the 200 μL dose will first receive half of the contents of one device using a dose divider and then 4 minutes later will receive the 2nd half by removing the dose divider. Subjects receiving the 400 μL dose will first receive the entire contents of one device and then 4 minutes later will receive the contents of a 2nd device.
  Other Names: Kovacaine Mist

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and safety of a nasal spray containing the anesthetic drug Tetracaine in combination with Oxymetazoline in healthy pediatric subjects.

DETAILED DESCRIPTION:
The purpose of this study is to determine the pharmacokinetics and safety of tetracaine, para- butylaminobenzoic acid (PBBA), and oxymetazoline after intranasal administration of the recommended, weight-based Phase 3 dose of Kovacaine Mist (Tetracaine Hydrochloride with Oxymetazoline Hydrochloride) to healthy pediatric subjects.

Kovacaine Mist is an anesthetic solution containing 3% tetracaine hydrochloride and 0.05% oxymetazoline hydrochloride. A single spray dose of 100 μL Kovacaine Mist contains 3 mg tetracaine HCl and 0.05 mg oxymetazoline HCl. A two-100 μL spray dose (a total of 200 μL) of Kovacaine Mist contains 6 mg tetracaine HCl and 0.1 mg oxymetazoline HCl. A two-200 μL spray dose (a total of 400 μL) of Kovacaine Mist contains 12 mg tetracaine HCl and 0.2 mg oxymetazoline HCl.

Kovacaine Mist will be administered based on the weight of the subject as summarized in the table below. Subjects weighing 10 to <20 kg will receive 1 intranasal spray of 100 μL of Kovacaine Mist at time D0. Subjects weighing 20 to <40 kg will receive 2 intranasal sprays of 100 μL (total dose 200 μL) administered 4 minutes apart at times D0 and D4. Subjects weighing 40 kg or more will receive 2 intranasal sprays of 200 μL (total dose 400 μL) administered 4 minutes apart at times D0 and D4.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 3-17 years of age inclusive.
* Sufficiently healthy as determined by the investigator to receive the test medications.
* Accompanied and/or represented by a parent or guardian able to comprehend and sign the informed consent document.
* Subject able to understand and provide assent to an age-appropriate subject assent form (as defined by local practice or regulation).
* Patient or parent/guardian able to communicate with the investigator and comply with the requirements of the protocol.
* Within the 10th and 90th percentiles for weight by age.
* Can breathe through both nostrils.
* Body mass index from 14 and 30 kg/m2 inclusive.

Exclusion Criteria:

* Any chronic or currently uncontrolled psychiatric, neurological, endocrine, pulmonary, cardiovascular, renal, gastrointestinal or hepatic disease or condition with manifestations that might confound interpretation of study results or make receipt of study medication a source of risk for adverse outcome.
* Inadequately controlled thyroid disease of any type.
* Has clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory evaluation during screening.
* Currently experiencing seasonal or perennial allergic rhinitis, recurrent nose-bleeds or asthma, or has a significant history of these conditions, in the opinion of the Investigator.
* Current, including the last 30 days, sinusitis or other upper respiratory infections, nasal congestion or use of a "sinus medication" within the 48 hours prior to anticipated study participation.
* Nasal polyps, significant nasal or sinus surgery or other abnormality that may interfere with the dose administration.
* History of allergy to or intolerance of tetracaine, oxymetazoline, benzyl alcohol, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreen).
* Use of a monoamine oxidase inhibitor within the 3 weeks preceding study entry.
* Nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females of child-bearing potential will be required to undergo urine testing at the baseline visit to rule out pregnancy.)
* Having received any investigational drug (including Kovacaine Mist) and/or participation in any clinical trial within 30 days of study participation.
* History of congenital or idiopathic methemoglobinemia.
* Anticipated need for use of oxymetazoline or phenylephrine nasal spray, nasal irrigation, or other nasal or oral decongestant on the day of the study procedure.
* Have a history of pseudocholinesterase deficiency or previous prolonged paralysis with succinylcholine or difficulty waking up from general anesthesia.
* Fever defined as body temperature ≥100.4 (38°C) on the day of and prior to study drug administration.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of tetracaine | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Time to Peak Plasma Concentration (Cmax) of tetracaine | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Terminal elimination rate constant (λz) of tetracaine | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Elimination half-life (t½) of tetracaine | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Area under the plasma concentration versus time curve (AUC) of tetracaine | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Peak Plasma Concentration (Cmax) of para- butylaminobenzoic acid (PBBA) | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Time to Peak Plasma Concentration (Cmax) of para- butylaminobenzoic acid (PBBA) | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Terminal elimination rate constant (λz) of para- butylaminobenzoic acid (PBBA) | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Elimination half-life (t½) of para- butylaminobenzoic acid (PBBA) | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Area under the plasma concentration versus time curve (AUC) of para- butylaminobenzoic acid (PBBA) | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Peak Plasma Concentration (Cmax) of oxymetazoline | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Time to Peak Plasma Concentration (Cmax) of oxymetazoline | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Terminal elimination rate constant (λz) of oxymetazoline | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Elimination half-life (t½) of oxymetazoline | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Area under the plasma concentration versus time curve (AUC) of oxymetazoline | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray

SECONDARY OUTCOMES:
Mean and Standard Deviation of Heart Rate | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Mean and Standard Deviation of Systolic Blood Pressure | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Mean and Standard Deviation of Diastolic Blood Pressure | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Mean and Standard Deviation of Temperature | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray
Mean and Standard Deviation of Oxygen Saturation | 0, 10, 30 minutes, and 1, 3, 6, 8, 9, 12, and 24 hours after completion of the last nasal spray

CONTACTS AND LOCATIONS:
Locations (1):
- AXIS Clinical Trials Research Center, Los Angeles, California, United States